CLINICAL TRIAL: NCT03433118
Title: A Feasibility Study of Acupuncture to Improve Quality of Life and Fatigue in Cancer Patients Undergoing Radiotherapy Treatment
Brief Title: Acupuncture in Cancer Patients Undergoing Radiotherapy Treatment
Acronym: ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal London Hospital for Integrated Medicine (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/0357
Record Dates: First submitted 2017-02-24; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Cancer
Keywords: fatigue; health-related quality of life
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT) comparing standard care against standard care with additional acupuncture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture administered by specially-trained therapeutic radiographers to patients attending the UCH radiotherapy department for radiotherapy intended to be curative of their cancer
  Interventions: Device: Acupuncture
- Standard care (No Intervention): Standard care for patients attending the UCH radiotherapy department for radiotherapy intended to be curative of their cancer

INTERVENTIONS:
Device: Acupuncture — Acupuncture administered by specially-trained therapeutic radiographers
  Arms: Acupuncture

SUMMARY:
Feasibility randomized controlled trial of standard care v standard care + acupuncture administered by specially-trained therapy radiographers in patients undergoing radiotherapy. It is a feasibility study to investigate all aspects of a future definitive randomized controlled trial, including statistical power calculation, hence there is no primary outcome or time point.

Mixed methods: literature review, model validity, training and mentoring of radiographers, processes, resources, interventions, procedures, patient clinical outcomes, patient and stakeholder qualitative outcomes

DETAILED DESCRIPTION:
The aim of the 'Acupuncture to improve quality of life and fatigue in cancer patients undergoing Radiotherapy Treatment' (ART) project is to investigate all aspects of the feasibility of undertaking clinical research on acupuncture with patients having radiotherapy at the University College Hospital (UCH) Cancer division.

The program includes an exploratory feasibility randomized controlled trial to investigate all aspects of a future definitive randomized controlled trial, including: organizational and procedural issues, patient group (including cancer diagnosis and stage), statistical power calculation, primary outcome measure and time point. It is NOT intended to deliver definitive results in terms of clinical outcomes.

ART aims to establish a platform for the investigation of integrating complementary therapy into cancer care, between the Royal London Hospital for Integrated Medicine (RLHIM) and the UCH cancer division. The development of a research project to investigate the use of acupuncture, a therapy not currently provided by the cancer division, to address the key concerns of cancer patients was the starting point. The intention is to evaluate the feasibility of such research, not to produce definitive results.

The greatest concerns of people with cancer include anxiety, fatigue, sleep problems and pain as a consequence of their disease and its treatment. Many patients find complementary therapies beneficial for these problems. UCH and RLHIM are both part of the University College London Hospital NHS Trust. The RLHIM is a specialist provider of complementary therapies, and offers treatment to cancer patients attending for radiotherapy and chemotherapy at UCH.

ART uses multiple methods, including a systematic review of the literature, model validity expert consensus, a novel therapy (acupuncture) and mode of delivery (specially trained health professionals already working in the radiotherapy department), and standard measures of outcome, culminating in a feasibility randomized controlled clinical trial.

The research program will evaluate all involved processes, resources, interventions and procedures. Outcomes measured included patient clinical outcomes, and the views of patients and stakeholders.

The research team comprises the Royal London Hospital for Integrated Medicine (RLHIM) research team, UCH Cancer Clinical Trials Unit (CCTU), a Steering Group including representatives of all interested parties including patients, an International Scientific Advisory Committee, an Acupuncture Expert Panel, with support from Quality Health Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Patients due to receive radical (curative) radiotherapy
* Patients of either gender and older than 16 years old.
* Patients with any cancer diagnosis.
* Patients willing to participate in the study and be randomised to one of the two treatment arms.
* Patients willing to attend at least 3 acupuncture treatments if assigned to the acupuncture intervention.
* Palliative patients.
* Patients unwilling to participate (for instance due to needle phobia).
* Patients currently receiving acupuncture.
* Patients with a platelet count <20 000mm.
* Patients with a white blood cell count <1000mm.
* Patients with severe clotting dysfunction or who bruise spontaneously.
* Patients unable to complete the questionnaires as judged by the investigators.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
EORTC QLQC-30 | Change from baseline (T0) to end of radiotherapy (3-8 weeks depending on tumor site and stage) (T2)
  EORTC QLQC-30: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30. A well-validated quality of life questionnaire for cancer patients focusing on functional assessment. It consists of nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. High internal consistency and construct validity have been demonstrated.

SECONDARY OUTCOMES:
MFI | Change from baseline (T0) to end of radiotherapy (3-8 weeks depending on tumor site and stage) (T2)
  Multidimensional Fatigue Inventory. A well-validated scale comprising 20 items measuring general fatigue including dimensions of physical and mental fatigue.
MSAS | Change from baseline (T0) to end of radiotherapy (3-8 weeks depending on tumor site and stage) (T2)
  Memorial Symptom Assessment Scale. A multidimensional scale which evaluates 32 physical and psychological symptoms associated with cancer and its treatment.
EQ-5D-5L | Change from baseline (T0) to end of radiotherapy (3-8 weeks depending on tumor site and stage) (T2)
  European Quality of Life 5 Dimensions 5 levels. A well-validated instrument which includes five indices to represent patients' Health Related Quality of Life: mobility; self-care; usual activities; pain/discomfort; anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Fisher, MD, Principal Investigator — Royal London Hospital for Integrated Medicine
Locations (1):
- University College London Hospitals Cancer Clinical Trials Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No